CLINICAL TRIAL: NCT00570765
Title: A Study of INT-747 (6-ECDCA) Monotherapy in Patients With Primary Biliary Cirrhosis
Brief Title: Study of INT-747 as Monotherapy in Participants With Primary Biliary Cirrhosis (PBC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 747-201; 2007-001424-12 (EudraCT Number)
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Liver Cirrhosis, Biliary
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DB OCA 10 mg (Experimental): OCA 10 mg for 3 months during the DB phase.
  Interventions: Drug: Obeticholic Acid (OCA)
- DB OCA 50 mg (Experimental): OCA 50 mg for 3 months during the DB phase.
  Interventions: Drug: Obeticholic Acid (OCA)
- DB OCA Placebo (Placebo Comparator): Matching placebo for 3 months during the DB phase.
  Interventions: Drug: Placebo
- LTSE OCA Total (Experimental): After completion of the 3-month DB phase, all eligible participants were offered the opportunity to enter an open-label LTSE for up to 96 months beginning at 10 mg OCA. Doses up to 50 mg daily were evaluated.
  Interventions: Drug: Obeticholic Acid (OCA)

INTERVENTIONS:
Drug: Placebo — Matching placebo tablets were administered orally once daily.
  Arms: DB OCA Placebo
Drug: Obeticholic Acid (OCA) — Starting dose of 10 or 50 mg administered orally once daily, followed by dose titration planned from 10 mg to 25 mg to 50 mg once daily, which could be modified for safety and tolerability issues or to achieve adequate therapeutic response.
  Other Names: INT-747; 6α-ethyl-chenodeoxycholic acid (6-ECDCA)
  Arms: DB OCA 10 mg; DB OCA 50 mg; LTSE OCA Total

SUMMARY:
The primary hypothesis was that obeticholic acid (OCA) will cause a reduction in alkaline phosphatase levels in PBC participants, over a 12-week treatment period, as compared to placebo.

DETAILED DESCRIPTION:
The study included 2 phases: a 3-month randomized, double-blind (DB), placebo-controlled, parallel group phase, followed by a long-term safety extension (LTSE). The planned duration of the LTSE phase was country-specific, ranging from 108 months to indefinitely. On-site visits occurred at least every 6 months.

Following completion of the 3-month DB phase, participants who continued to meet protocol requirements were given the opportunity to enroll in the LTSE phase of the study at selected study sites. The participants who enrolled in the LTSE phase started OCA administration, from a starting dose (10 or 50 milligrams [mg]) based on the dose of OCA or placebo received in the DB phase or on the timing of entry into the LTSE phase.

Because the LTSE phase was not planned in the original study design, participants had varied gaps between the end of the DB phase and the start of the LTSE phase. Moreover, some participants initiated ursodeoxycholic acid during the course of that break.

ELIGIBILITY:
Inclusion Criteria:

* Female participants must be postmenopausal, surgically sterile, or if premenopausal, be prepared to use 1 effective method of contraception with all sexual partners during the study and for 14 days after the end of dosing.
* Male participants must be prepared to use 1 effective method of contraception with all sexual partners during the study during the study unless they had a prior vasectomy.
* Proven or likely PBC, as demonstrated by the participant presenting with at least 2 of the following 3 diagnostic factors:
* History of increased alkaline phosphatase (ALP) levels for at least 6 months;
* Positive antimitochondrial antibody titer (>1:40 titer on immunofluorescence or M2 positive by enzyme-linked immunosorbent assay) or PBC-specific antinuclear antibodies (antinuclear dot and nuclear rim positive);
* Liver biopsy consistent with PBC
* Screening ALP level between 1.5 and 10 × upper limit of normal (ULN).

Exclusion Criteria:

* Administration of the following drugs at any time during the 3 months prior to screening for the study: ursodeoxycholic acid, colchicine, methotrexate, azathioprine, or systemic corticosteroids.
* Screening conjugated (direct) bilirubin >2 × ULN.
* Screening alanine aminotransferase or aspartate aminotransferase >5 × ULN.
* Screening serum creatinine >133 micromoles/liter (1.5 mg/deciliter).

History or presence of hepatic decompensation (for example, variceal bleeds, encephalopathy, or poorly controlled ascites).

* History or presence of other concomitant liver diseases including hepatitis due to hepatitis B or C virus infection, primary sclerosing cholangitis, alcoholic liver disease, definite autoimmune liver disease or biopsy proven nonalcoholic steatohepatitis.
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-01-17 (Actual); Primary Completion 2010-09-21 (Actual); Study Completion 2017-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Weyer, MD, Study Chair — Intercept Pharmaceuticals, Inc.
Locations (21):
- United States (4):
  - Henry Ford, Detroit, Michigan
  - Baylor College of Medicine, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Karls-Franzens University, Graz, Austria
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - University of Toronto, Toronto, Ontario
  - Centre de Recherche du CHUM / University of Montreal, Montreal, Quebec
- France (2):
  - Hopital de l'Hotel Dieu, Lyon
  - Hopital Saint-Antoine, Paris
- Germany (4):
  - Johann Wolfgang Goethe University, Frankfurt
  - University Medical Centre Hamburg-Eppendorf, Hamburg
  - Medical School of Hannover, Hanover
  - University of Munich, Munich
- Hospital Clinic i Provincial, Barcelona, Spain
- United Kingdom (6):
  - Queen Elizabeth Medical Center, Edgbaston, Birmingham
  - Royal Free Hospital, Hampstead, London
  - John Radcliffe Hospital, Headington, Oxford
  - Royal Infirmary, Edinburgh
  - Sunderland Research Ethics Committee, Jarrow
  - University Upon Tyne/Newcastle, Newcastle upon Tyne

REFERENCES:
- [Background] Kowdley KV, Luketic V, Chapman R, Hirschfield GM, Poupon R, Schramm C, Vincent C, Rust C, Pares A, Mason A, Marschall HU, Shapiro D, Adorini L, Sciacca C, Beecher-Jones T, Bohm O, Pencek R, Jones D; Obeticholic Acid PBC Monotherapy Study Group. A randomized trial of obeticholic acid monotherapy in patients with primary biliary cholangitis. Hepatology. 2018 May;67(5):1890-1902. doi: 10.1002/hep.29569. Epub 2018 Jan 29. PMID 29023915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started Dec. 2007 and completed June 2010. Due to positive Phase 2 data in another study (NCT00550862), power calculations were revised and recruitment ended early. Eligible participants who received treatment in the double-blind (DB) phase could continue receiving obeticholic acid (OCA) in the long-term safety extension (LTSE) phase.
Pre-assignment Details: Screening interim allowed for pre-randomization eligibility assessment of 1 to 4 weeks. Other than 3-month (pre-Screening) washout for ursodeoxycholic acid and other medications, no washout or run-in period was defined between Screening and Randomization. During LTSE, OCA dosing (milligrams [mg]) remained oral once daily.
Period: DB Phase
Arm/Group | DB OCA 10 mg | DB OCA 50 mg | DB OCA Placebo | LTSE OCA Total
Started | 20 | 16 | 24 | 0
Received at Least 1 Dose of Study Drug | 20 | 16 | 23 | 0
Safety Population | 20 | 16 | 23 | 0
Completed | 16 | 9 | 23 | 0
Not Completed | 4 | 7 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 6 | 0 | 0
Not completed — Did Not Receive Study Drug | 0 | 0 | 1 | 0
Period: LTSE Phase
Arm/Group | DB OCA 10 mg | DB OCA 50 mg | DB OCA Placebo | LTSE OCA Total
Started | 0 (Eligible participants who completed the DB phase enrolled in the LTSE phase.) | 0 (Eligible participants who completed the DB phase enrolled in the LTSE phase.) | 0 (Eligible participants who completed the DB phase enrolled in the LTSE phase.) | 28 (Eligible participants who completed the DB phase enrolled in the LTSE phase.)
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 28
Safety Population | 0 | 0 | 0 | 28
Completed | 0 | 0 | 0 | 16
Not Completed | 0 | 0 | 0 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 7
Not completed — Physician Decision | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Safety Population: all randomized participants who received at least 1 dose of investigational product based on the treatment group assignment and had at least 1 post-treatment safety assessment.
Groups:
- DB OCA 10 mg: OCA 10 mg for 3 months during the DB phase. After completion of the 3-month DB phase, all eligible participants were offered the opportunity to enter an open-label LTSE for up to 96 months beginning at 10 mg OCA. Doses up to 50 mg daily were evaluated.
- DB OCA 50 mg: OCA 50 mg for 3 months during the DB phase. After completion of the 3-month DB phase, all eligible participants were offered the opportunity to enter an open-label LTSE for up to 96 months beginning at 10 mg OCA. Doses up to 50 mg daily were evaluated.
- DB OCA Placebo: Matching placebo for 3 months during the DB phase. After completion of the 3-month DB phase, all eligible participants were offered the opportunity to enter an open-label LTSE for up to 96 months beginning at 10 mg OCA. Doses up to 50 mg daily were evaluated.
- Total: Total of all reporting groups
Arm/Group | DB OCA 10 mg | DB OCA 50 mg | DB OCA Placebo | Total
Number analyzed (Participants) | 20 | 16 | 23 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 18 | 49
  >=65 years | 4 | 1 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.9) | 54.1 (7.3) | 55.3 (10.0) | 54.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 20 | 50
  Male | 6 | 0 | 3 | 9
Region of Enrollment [Number; unit: participants]
  France | 2 | 1 | 1 | 4
  United States | 4 | 5 | 8 | 17
  Canada | 3 | 2 | 4 | 9
  Spain | 0 | 1 | 1 | 2
  Germany | 4 | 1 | 3 | 8
  United Kingdom | 7 | 6 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: DB Phase: Mean Percent Change In Serum Alkaline Phosphatase (ALP) From Baseline To Day 85
Description: The percent change in serum ALP from baseline to Day 85 is reported. The baseline value used was the mean of the pretreatment Screening and Day 0 evaluations.
Time Frame: Baseline, Day 85
Population: Intention-to-treat (ITT): participants randomized to receive investigational product regardless of their actual treatment status.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DB OCA 10 mg | DB OCA 50 mg | DB OCA Placebo
Number analyzed (Participants) | 20 | 16 | 23
Percent change | -44.5 (24.4) | -37.6 (21.0) | 0.4 (15.3)
Statistical Analysis 1: Comparison: DB OCA 10 mg vs DB OCA 50 mg vs DB OCA Placebo; Hierarchical testing strategy was proposed to account for multiple comparisons. Statistical significance was evaluated as follows: if statistical significance at alpha=0.05 is shown for the 10 mg OCA versus placebo, then the statistical significance at alpha=0.05 for the 50 mg OCA versus placebo was evaluated. If no statistical significance was shown at alpha=0.05 at the first step, then the subsequent comparison was not considered statistically significant; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Treatment arms compared using 2-sided Wilcoxon-Mann-Whitney test at 5% significance level. Treatment groups were pairwise compared versus placebo

2. Secondary Outcome: DB Phase: Mean Percent Change In Gamma-glutamyl Transferase (GGT) From Baseline To Day 85
Description: As a marker of hepatocellular injury and liver function, the percent change in GGT from baseline to Day 85 is reported.
Time Frame: Baseline, Day 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DB OCA 10 mg | DB OCA 50 mg | DB OCA Placebo
Number analyzed (Participants) | 19 | 15 | 22
Percent change | -73 (18) | -65 (25) | -3 (22)
Statistical Analysis 1: Comparison: DB OCA 10 mg vs DB OCA 50 mg vs DB OCA Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: DB Phase: Mean Percent Change In Alanine Transaminase (ALT) From Baseline To Day 85
Description: As a marker of hepatocellular injury and liver function, the percent change in ALT from baseline to Day 85 is reported.
Time Frame: Baseline, Day 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DB OCA 10 mg | DB OCA 50 mg | DB OCA Placebo
Number analyzed (Participants) | 19 | 15 | 22
Percent change | -37 (35) | -35 (25) | -4 (40)
Statistical Analysis 1: Comparison: DB OCA 10 mg vs DB OCA 50 mg vs DB OCA Placebo; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney); Tx arms will be compared using the 2-sided Wilcoxon-Mann-Whitney test, at 5% significance level. Tx groups will be pairwise compared vs. placebo

4. Secondary Outcome: DB: Plasma Trough Concentrations Of OCA And Its Major, Known Metabolites
Time Frame: 12 weeks
Population: OCA and its conjugates were quantified by an assay using an extended and improved protocol initially described in peer reviewed literature. The assay was not validated when the study was conducted. A validated assay was established using plasma after the study. But because only serum samples, not plasma samples, were acquired in the study, the levels of OCA and its conjugates were not summarized in the clinical study report, and thus, not used to draw conclusions on exposure.
Arm/Group | DB OCA 10 mg | DB OCA 50 mg | DB OCA Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: DB Phase: Mean Percent Change In Conjugated Bilirubin From Baseline To Day 85
Description: As a marker of hepatocellular injury and liver function, the percent change in conjugated bilirubin from baseline to Day 85 is reported.
Time Frame: Baseline, Day 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | DB OCA 10 mg | DB OCA 50 mg | DB OCA Placebo
Number analyzed (Participants) | 18 | 15 | 22
Percent Change | 0.7 (67.3) | -1.7 (39.9) | 30.3 (69.8)

6. Secondary Outcome: LTSE Phase: Median Percent Change In Serum ALP From Baseline To Month 24, Month 48, Month 72, And Last Available Visit
Description: The percent change in serum ALP from baseline to the last available visit is reported. The DB baseline value was used as the baseline.
Time Frame: Baseline (DB), Month 24, Month 48, Month 72, Last Available Visit (up to 96 months)
Population: Safety Population: participants who received at least 1 dose of open-label investigational product during the LTSE phase.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 28
Percent Change
  Month 24: number analyzed (Participants) | 23
  Month 24 | -43.1 [-61.3 to -20.2]
  Month 48: number analyzed (Participants) | 19
  Month 48 | -44.4 [-65.5 to -18.6]
  Month 72: number analyzed (Participants) | 17
  Month 72 | -33.4 [-64.5 to -17.9]
  Last Available Visit | -31.8 [-57.5 to -14.0]

7. Secondary Outcome: LTSE Phase: Mean Percent Change In Serum ALP From Baseline To Month 24, Month 48, Month 72, And Last Available Visit
Description: as for outcome 6
Time Frame: Baseline (DB), Month 24, Month 48, Month 72, Last Available Visit (up to 96 months)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 28
Percent Change
  Month 24: number analyzed (Participants) | 23
  Month 24 | -38.8 (29.7)
  Month 48: number analyzed (Participants) | 19
  Month 48 | -39.3 (36.6)
  Month 72: number analyzed (Participants) | 17
  Month 72 | -31.7 (57.3)
  Last Available Visit | -30.4 (36.6)

8. Secondary Outcome: LTSE: Median Percent Change In GGT From Baseline To Last Available Visit
Description: As a marker of hepatocellular injury and liver function, the percent change in GGT from baseline to the last available visit is reported. The DB baseline value was used as the baseline.
Time Frame: Baseline (DB), Last Available Visit (up to 96 months)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 28
Percent Change | -71.1 [-84.3 to -33.8]

9. Secondary Outcome: LTSE: Mean Percent Change In GGT From Baseline To Last Available Visit
Description: as for outcome 8
Time Frame: Baseline (DB), Last Available Visit (up to 96 months)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 28
Percent Change | -55.6 (41.4)

10. Secondary Outcome: LTSE: Median Percent Change In ALT From Baseline To Last Available Visit
Description: As a marker of hepatocellular injury and liver function, the percent change in ALT from baseline to the last available visit is reported. The DB baseline value was used as the baseline.
Time Frame: Baseline (DB), Last Available Visit (up to 96 months)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 28
Percent Change | -52.2 [-68.4 to -11.6]

11. Secondary Outcome: LTSE: Mean Percent Change In ALT From Baseline To Last Available Visit
Description: as for outcome 10
Time Frame: Baseline (DB), Last Available Visit (up to 96 months)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 28
Percent Change | -39.6 (42.8)

12. Secondary Outcome: LTSE: Median Percent Change In Conjugated Bilirubin From Baseline To Last Available Visit
Description: As a marker of hepatocellular injury and liver function, the percent change in conjugated bilirubin from baseline to the last available visit is reported. The DB baseline value was used as the baseline.
Time Frame: Baseline (DB), Last Available Visit (up to 96 months)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Percent Change
Groups:
- LTSE OCA Total: After completion of the 3-month DB phase, all eligible participants were offered the opportunity to enter an open-label LTSE for up to 96 months beginning at 10 mg OCA (PO QD). Doses up to 50 mg daily were evaluated.
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 28
Percent Change | 33.3 [-11.1 to 100.0]

13. Secondary Outcome: LTSE: Mean Percent Change In Conjugated Bilirubin From Baseline To Last Available Visit
Description: as for outcome 12
Time Frame: Baseline (DB), Last Available Visit (up to 96 months)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 28
Percent Change | 57.8 (103.0)

14. Secondary Outcome: LTSE: Median Percent Change In Total Bilirubin From Baseline To Last Available Visit
Description: As a marker of hepatocellular injury and liver function, the percent change in total bilirubin from baseline to the last available visit is reported. The DB baseline value was used as the baseline.
Time Frame: Baseline (DB), Last Available Visit (up to 96 months)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 28
Percent Change | 5.2 [-21.4 to 25.2]

15. Secondary Outcome: LTSE: Mean Percent Change In Total Bilirubin From Baseline To Last Available Visit
Description: as for outcome 14
Time Frame: Baseline (DB), Last Available Visit (up to 96 months)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | LTSE OCA Total
Number analyzed (Participants) | 28
Percent Change | 2.2 (35.1)

ADVERSE EVENTS:
Time Frame: DB Phase: Adverse events were collected starting when the participant took the first dose of study medication (following Day 0) and during study participation, through the follow-up visit at Month 3. LSTE Phase: Baseline (DB Month 3) up to 96 months.
Arm/Group | DB OCA 10 mg | DB OCA 50 mg | DB OCA Placebo | LTSE OCA Total
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/16 | 1/23 | 9/28
Other Adverse Events (participants affected / at risk) | 18/20 | 15/16 | 19/23 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DB OCA 10 mg (N=20) | DB OCA 50 mg (N=16) | DB OCA Placebo (N=23) | LTSE OCA Total (N=28)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant hospitalized due to hypersensitivity to opioids.
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 0/14 (0) | 0 (0) | 0/20 (0) | 1/23 (1) — This adverse event affected only female participants.
Cystocele (Reproductive system and breast disorders) | 0/14 (0) | 0 (0) | 0/20 (0) | 1/23 (1) — This adverse event affected only female participants.
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.99% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DB OCA 10 mg (N=20) | DB OCA 50 mg (N=16) | DB OCA Placebo (N=23) | LTSE OCA Total (N=28)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (24) | 15 (22) | 7 (11) | 25 (107)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 8 (12)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 4 (5) | 5 (5)
Fatigue (General disorders) | 0 (0) | 1 (1) | 3 (3) | 14 (16)
Headache (Nervous system disorders) | 4 (5) | 2 (3) | 5 (6) | 8 (12)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (7)
Insomnia (Psychiatric disorders) | 1 (2) | 2 (2) | 1 (1) | 5 (6)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 3 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (5) | 11 (19)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 5 (9)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Iritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 9 (11)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (10)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 6 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (7)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 5 (5)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Faeces pale (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (11)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 6 (11)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 9 (11)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 4 (6)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 4 (6)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cells urine (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 13 (33)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (8)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (6)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Facial neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irregular sleep phase (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 1/14 (1) | 0 (0) | 0/20 (0) | 1/23 (2) — This adverse event affected only female participants.
Ovarian cyst (Reproductive system and breast disorders) | 0/14 (0) | 0 (0) | 0/20 (0) | 2/23 (2) — This adverse event affected only female participants.
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1/14 (1) | 0 (0) | 0/20 (0) | 0/23 (0) — This adverse event affected only female participants.
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Spider naevus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of the study include the use of ursodeoxycholic acid that disallowed meeting key inclusion/exclusion criteria, a short double-blind phase, and the reason participants were not receiving ursodeoxycholic acid at baseline was not captured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per protocol, Intercept retains ownership of the study data. Proposed publications based on the study shall be approved prior to submission for publications and will not be unreasonably withheld.